CLINICAL TRIAL: NCT05251194
Title: The Effect of McGrath Video Laryngoscope on the Glottic View at Thyroid Surgery Position in Tracheal Intubation
Brief Title: The Effect of McGrath Video Laryngoscope on the Glottic View at Thyroid Surgery Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2022-3
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Thyroid Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video laryngoscope at thyroid surgical position (Experimental): After induction of anesthesia and muscle relaxation, the patient will be positioned with a standard pillow to exposure neck for thyroid surgery (thyroid surgical position). Then, tracheal intubation will be performed with a McGrath video laryngoscope. During laryngoscopy with the McGrath video laryngoscope, the intubation practitioner will record the modified Cormack-Lehane grade and the percentage of glottic opening (POGO) score when it is assumed that a direct laryngoscope is used and when using the video laryngoscope, respectively.
  Next, the intubation practitioner will perform tracheal intubation with it.
  Interventions: Device: video laryngoscope at thyroid surgical position

INTERVENTIONS:
Device: video laryngoscope at thyroid surgical position — After induction of anesthesia and muscle relaxation, the patient will be positioned with a standard pillow to exposure neck for thyroid surgery (thyroid surgical position). Then, tracheal intubation will be performed with a McGrath video laryngoscope. During laryngoscopy with the McGrath video laryngoscope, the intubation practitioner will record the modified Cormack-Lehane grade and the percentage of glottic opening (POGO) score when it is assumed that a direct laryngoscope is used and when using the video laryngoscope, respectively.

SUMMARY:
For thyroid surgery, the special body position (thyroid surgical position) to exposure the patient's neck should be needed. For intraoperative neuromonitoring (IONM) in thyroid surgery, the tube should be placed at a specific position. A video laryngoscope can have advantages in tracheal intubation on thyroid surgical position for thyroid surgery. The purpose of the study is to investigate the effect of McGrath video laryngoscope on the glottic view when tracheal intubation is performed at the thyroid surgical position.

DETAILED DESCRIPTION:
For thyroid surgery, the special body position (thyroid surgical position) to exposure the patient's neck should be needed. Meanwhile, the tracheal tube can be moved in the trachea from the supine position to thyroid surgical position if tracheal intubation is performed at the supine position. For intraoperative neuromonitoring (IONM) in thyroid surgery, the electrode of the tracheal tube must be placed at a specific position, that is between the vocal cords. To perform initially tracheal intubation on the thyroid surgical position, therefore, can have advantage in terms of stability of tube position in the trachea without displacement by body position change. However, tracheal intubation on thyroid surgical position might be hard in terms of obtaining a good glottic view. It is well known that video laryngoscopes can improve the glottic view. Therefore, a video laryngoscope can have advantages in tracheal intubation on thyroid surgical position for thyroid surgery in obtaining the good glottic view as well as minimal displacement of the tracheal tube because there is no need to change the patient's position. The purpose of the study is to investigate the effect of McGrath video laryngoscope on the glottic view when tracheal intubation is performed at the thyroid surgical position.

ELIGIBILITY:
Inclusion Criteria:

* patients schedule to thyroid surgery

Exclusion Criteria:

* disagree to participate
* patients with weak teeth

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
direct modified Cormack-Lehane grade without external manipulation | at tracheal intubation
  During laryngoscopy, the modified Cormack-Lehane grade without external manipulation as if the laryngoscope is assumed as a direct laryngoscope
direct percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) without external manipulation | at tracheal intubation
  During laryngoscopy, the percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) without external manipulation as if the laryngoscope is assumed as a direct laryngoscope
video modified Cormack-Lehane grade without external manipulation | at tracheal intubation
  During laryngoscopy, the modified Cormack-Lehane grade without external manipulation as if the laryngoscope is used as a video laryngoscope
video percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) without external manipulation | at tracheal intubation
  During laryngoscopy, the percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) without external manipulation as if the laryngoscope is used as a video laryngoscope
direct modified Cormack-Lehane grade with external manipulation | at tracheal intubation
  During laryngoscopy, the modified Cormack-Lehane grade with external manipulation as if the laryngoscope is assumed as a direct laryngoscope
direct percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) with external manipulation | at tracheal intubation
  During laryngoscopy, the percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) with external manipulation as if the laryngoscope is assumed as a direct laryngoscope
video modified Cormack-Lehane grade with external manipulation | at tracheal intubation
  During laryngoscopy, the modified Cormack-Lehane grade with external manipulation as if the laryngoscope is used as a video laryngoscope
video percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) with external manipulation | at tracheal intubation
  During laryngoscopy, the percentage of glottic opening score (POGO score: 0 - 100, 100 means full visualization of vocal cords) with external manipulation as if the laryngoscope is used as a video laryngoscope

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, MD.PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea